CLINICAL TRIAL: NCT00369668
Title: Subacute Stroke Recovery (Upper Extremity Motor Function): Bimanual Coordination Training
Brief Title: Post Stroke Hand Functions: Bilateral Movements and Electrical Stimulation Treatments
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00061194
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Results first posted 2012-05-11 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-04

CONDITIONS: Cerebrovascular Accident; Hemiplegia
Keywords: Rehabilitation; Physical Therapy Techniques; Occupational Therapy; Upper Extremity; Motor skills
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Intensity (Experimental): Bilateral training moving both arms coupled with neuromuscular electrical stimulation; four 90-minute sessions/week for 2 weeks.
  Interventions: Behavioral: Bilateral movements and neuromuscular electrical stimulation
- Low Intensity (Active Comparator): Bilateral training moving both arms coupled with neuromuscular electrical stimulation; two 90-minute sessions/week for 2 weeks.
  Interventions: Behavioral: Bilateral movements and neuromuscular electrical stimulation
- Control (Active Comparator): Bilateral training moving both arms coupled with sham neuromuscular electrical stimulation
  Interventions: Behavioral: Bilateral movements and sham electrical stimulation

INTERVENTIONS:
Behavioral: Bilateral movements and neuromuscular electrical stimulation — Participants practice moving their paretic arm at the same time as they move their non-paretic arm in the same movement patterns. Neuromuscular electrical stimulation triggered by the participants' own contracting muscles is provided to the paretic arm during the movements. Training period was 4 times per week for 2 weeks.
  Other Names: functional electrical stimulation
  Arms: High Intensity
Behavioral: Bilateral movements and neuromuscular electrical stimulation — Participants practice moving both their paretic and non-paretic arms at the same time in the same movement patterns. Neuromuscular electrical stimulation triggered by the participants' own contracting muscles is provided to the paretic arm during the movements. Training period was 2 times per week for 2 weeks.
  Other Names: functional electrical stimulation
  Arms: Low Intensity
Behavioral: Bilateral movements and sham electrical stimulation — Participants practice moving both their paretic and non-paretic arms at the same time in the same movement patterns. Sham electrical stimulation (low level electrical stimulation that can be felt but is insufficient to trigger a muscle contraction) is provided to the paretic arm during the movement. Training period was 2 times per week for 2 weeks.
  Other Names: functional electrical stimulation - sham
  Arms: Control

SUMMARY:
The purpose of this study was to determine the effect of two amounts of treatment therapy on post stroke motor recovery in the arms. The therapy is bilateral movement training combined with electrical stimulation on the impaired limb.

DETAILED DESCRIPTION:
Intense movement training (practice) with the affected arm after stroke has the potential to improve upper extremity (UE) function resulting from neuroplasticity changes in the motor cortex. However, the necessary and sufficient parameters of this therapy in humans have not been fully investigated. Delineation of the most efficacious and efficient therapy for promoting UE recovery post-stroke is necessary before effective clinical implementation of this therapy. The current compared the effects on motor function impairments for three bilateral movement groups involving two doses of treatment (i.e., bilateral training coupled with neuromuscular electrical stimulation) and a sham control. During the subacute recovery phase (3 - 6 months), patients who meet motor capabilities criteria will be randomly assigned to one of three groups: (a) low intensity: 90 minutes/session, 2 sessions/week 2 weeks; bilateral movement training coupled with active neuromuscular stimulation on the impaired wrist/fingers; (b) high intensity: 90 minutes/session, 4 sessions/week for 2 weeks; bilateral movement training coupled with active stimulation on the impaired wrist/finger extensors; and (c) control group (sham active stimulation). Patients' UE motor capabilities were assessed before treatment therapy began (pretest) and within the first week after the treatment therapy ended (posttest).

ELIGIBILITY:
Inclusion Criteria:

* an ability to complete 10º of wrist or finger extension from a 60 - 65 º flexed position
* score less than a 56 on the UE subscale of the Fugl-Meyer Assessment
* an ability to voluntarily activate slight movements in the wrist and fingers so that the EMG activity reaches a minimal level on the microprocessor for electrical stimulation to be activated
* unilateral, first stroke of ischemic or hemorrhagic origin in the carotid artery distribution
* free of major post stroke complications
* able to attend therapy 2 days/week or 4 days/week for 2 weeks
* score at least a 16 on the Mini Mental Status Examination
* able to discriminate sharp from dull and light touch using traditional sensation tests.

Exclusion Criteria:

* hemiparetic arm is insensate
* motor impairments from stroke on opposite side of body
* pre-existing neurological disorders such as Parkinson's disease, Multiple Sclerosis, or dementia
* Legal blindness or severe visual impairment; 5) Life expectancy less than one year
* Severe arthritis or orthopedic problems that limit passive ranges of motion of upper extremity (passive finger extension < 40º; passive wrist extension < 40º; passive elbow extension <40º; shoulder flexion/abduction < 80º)
* History of sustained alcoholism or drug abuse in the last six months
* Has pacemaker or other implanted device
* pregnant

Ages: 44 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James H. Cauraugh, Ph.D., Principal Investigator — University of Florida
Locations (1):
- Motor Behavior Laboratory, University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Cauraugh JH, Coombes SA, Lodha N, Naik SK, Summers JJ. Upper extremity improvements in chronic stroke: coupled bilateral load training. Restor Neurol Neurosci. 2009;27(1):17-25. doi: 10.3233/RNN-2009-0455. PMID 19164850
- [Result] Cauraugh JH, Kim SB. Stroke motor recovery: active neuromuscular stimulation and repetitive practice schedules. J Neurol Neurosurg Psychiatry. 2003 Nov;74(11):1562-6. doi: 10.1136/jnnp.74.11.1562. PMID 14617717
- [Result] Cauraugh JH, Kim S. Two coupled motor recovery protocols are better than one: electromyogram-triggered neuromuscular stimulation and bilateral movements. Stroke. 2002 Jun;33(6):1589-94. doi: 10.1161/01.str.0000016926.77114.a6. PMID 12052996
- [Result] Cauraugh JH, Kim SB. Chronic stroke motor recovery: duration of active neuromuscular stimulation. J Neurol Sci. 2003 Nov 15;215(1-2):13-9. doi: 10.1016/s0022-510x(03)00169-2. PMID 14568122
- [Result] Richards LG, Stewart KC, Woodbury ML, Senesac C, Cauraugh JH. Movement-dependent stroke recovery: a systematic review and meta-analysis of TMS and fMRI evidence. Neuropsychologia. 2008 Jan 15;46(1):3-11. doi: 10.1016/j.neuropsychologia.2007.08.013. Epub 2007 Aug 24. PMID 17904594
- [Result] Lodha N, Naik SK, Coombes SA, Cauraugh JH. Force control and degree of motor impairments in chronic stroke. Clin Neurophysiol. 2010 Nov;121(11):1952-61. doi: 10.1016/j.clinph.2010.04.005. PMID 20435515
- [Result] Naik SK, Patten C, Lodha N, Coombes SA, Cauraugh JH. Force control deficits in chronic stroke: grip formation and release phases. Exp Brain Res. 2011 May;211(1):1-15. doi: 10.1007/s00221-011-2637-8. Epub 2011 Mar 30. PMID 21448576
- [Result] Cauraugh JH, Lodha N, Naik SK, Summers JJ. Bilateral movement training and stroke motor recovery progress: a structured review and meta-analysis. Hum Mov Sci. 2010 Oct;29(5):853-70. doi: 10.1016/j.humov.2009.09.004. Epub 2009 Nov 18. PMID 19926154
- [Derived] Clark B, Whitall J, Kwakkel G, Mehrholz J, Ewings S, Burridge J. The effect of time spent in rehabilitation on activity limitation and impairment after stroke. Cochrane Database Syst Rev. 2021 Oct 25;10(10):CD012612. doi: 10.1002/14651858.CD012612.pub2. PMID 34695300

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Started August 2006 and ended June 2009
Pre-assignment Details: Inability to voluntarily execute 10 degrees of wrist/finger extension from a 60-65 degrees flexed position.
Period: Overall Study
Arm/Group | High Intensity | Low Intensity | Control
Started | 10 (Original number of participants to be recruited for each group.) | 10 | 10
Completed | 6 | 5 | 3
Not Completed | 4 | 5 | 7
Not completed — Lack of Efficacy | 4 | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Intensity | Low Intensity | Control | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 5 | 12
  >=65 years | 6 | 7 | 5 | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 65.3 (8.1) | 67.2 (6.8) | 61.8 (2.6) | 65.2 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 5 | 17
  Male | 4 | 4 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Box and Block Test; Data Collected = Number of Blocks Moved
Description: A 60 second timed hand/arm manipulation test in which participants reach, grasp, lift, and release a 1" x 1" block of wood. They must lift a block from one side of a box, carry it over a low barrier and release the block into the other side of the box.
Time Frame: Baseline/pretest; posttest given between days 17-22 (posttest days 3 -8)
Population: All participants who completed the bilateral training protocols were submitted to statistical analysis. Data for all participants were collected twice: (a) baseline/pretest: before treatment and (b) posttest: after treatment.
Measure: Mean (Standard Deviation); unit: Blocks
Arm/Group | High Intensity | Low Intensity | Control
Number analyzed (Participants) | 6 | 5 | 3
Blocks
  Baseline/Pretest | 24.5 (22.1) | 24.6 (12.7) | 40 (27.1)
  Posttest | 27.5 (21.7) | 31.8 (12.6) | 42 (26.5)
Statistical Analysis 1: Comparison: High Intensity vs Low Intensity vs Control; Group by Test Session ANOVA with repeated measures on second factor; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Greenhouse-Geisser degrees of freedom adjustment was not necessary; Mean Difference (Final Values) = 30, 95% CI 2-sided [22.5 to 37.4], Standard Error of Mean 3.65

2. Primary Outcome: Fugl-Meyer Upper Extremity Motor Test
Description: FM motor test assesses functional impairments post stroke as participants attempt various movements from daily activities. Minimum score = 0; maximum score = 66; lower scores indicate more impairments and higher scores indicate less impairments.
Time Frame: Baseline/pretest; posttest given between days 17-22 (posttest days 3 -8)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- High Intensity: Bilateral movements coupled with neuromuscular electrical stimulation. Four times per week for two weeks.
- Low Intensity: Bilateral movements coupled with neuromuscular electrical stimulation. Two times per week for two weeks.
- Control: Bilateral movements coupled with sham neuromuscular electrical stimulation. Two times per week for two weeks.
Arm/Group | High Intensity | Low Intensity | Control
Number analyzed (Participants) | 6 | 5 | 3
units on a scale
  Baseline/Pretest | 39 (19.8) | 41 (16.3) | 53 (9.7)
  Posttest | 42 (17.1) | 45 (15.6) | 56 (6.9)

3. Primary Outcome: Fractionated Reaction Time
Description: Premotor reaction times in milliseconds were recorded for the impaired arm of each participant in the three intervention (arm) groups. Premotor reaction time represents central processes. Lower times are faster reaction times, indicating less time to initiate a movement.
Time Frame: Baseline/pretest; posttest given between days 17-22 (posttest days 3-8)
Population: All participants who completed the bilateral training protocols were submitted to statistical analysis. Premotor reaction data for all participants were collected twice: (a) baseline/pretest: before treatment and (b) posttest: after treatment.
Measure: Median (Standard Error); unit: milliseconds
Arm/Group | High Intensity | Low Intensity | Control
Number analyzed (Participants) | 6 | 5 | 3
milliseconds
  Baseline/Pretest | 179 (27.1) | 225 (19.3) | 135 (5.6)
  Posttest | 170 (22.8) | 241 (23.4) | 161 (5.4)

ADVERSE EVENTS:
Time Frame: 2 years, 10 months
Arm/Group | High Intensity | Low Intensity | Control
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No